CLINICAL TRIAL: NCT06658808
Title: Efficacy-Implementation Study for Promoting Community Conversations About Research to End Suicide (PC CARES) in Rural Alaska
Brief Title: Efficacy-Implementation Study for PC CARES in Rural Alaska
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Yukon Kuskokwim Health Corporation (Other); Norton Sound Health Corporation (Other); Maniilaq Association (Unknown); University of Alaska Fairbanks (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Wexler, Research Professor, Research Center for Group Dynamics, Institute for Social Research and Professor of Social Work, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00247458; 1R01MH136768-01 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Suicide Prevention
Keywords: Suicide Prevention; Alaska Native; Community Intervention; Community-Based Participatory Research
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The study will have a stepped wedge design with 3 cycles of implementation (in successive years) across 9-12 villages total, depending on need and feasibility to achieve our needs. In each village, we will collect baseline data and follow-up data on knowledge, attitudes, and behavior related to suicide prevention from participants and non-participants. Participants will also provide data on these topics after each learning circle they attend and non-participants will be given a monthly survey each month for 5 months as the learning circles occur. Intervention participants will be self-selecting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PC CARES Intervention (Experimental): PC CARES Intervention Participants will attend 1-5 sessions of the PC CARES curriculum, either virtually or in-person. Investigators will collect data from this group at baseline, after each session they attend, and at follow-up.
  Interventions: Behavioral: Promoting Community Conversations About Research to End Suicide
- No Intervention (No Intervention): This group will not attend the PC CARES sessions. Investigators will collect data from adults and youth at baseline, at 5 monthly timepoints as learning circles are being conducted in the community, and at follow-up (after 1 month and 6 months).

INTERVENTIONS:
Behavioral: Promoting Community Conversations About Research to End Suicide — Promoting Community Conversations About Research to End Suicide (PC CARES) trains local community health workers to facilitate a series of five 3-hour Learning Circles (LCs) over ~6 months to develop a 'community of practice' (CoP), whereby trusted adults of youth (a) learn about SPBPs; (b) tailor the SPBPs to their culture and community; (c) build cross-sector relationships (parents, teachers, etc.), and (d) do more to prevent suicide. Each session shares evidence-based, actionable ways to enhance social support, reduce harm/risk, and promote help seeking, which participants adapt and apply in their daily interactions with youth.
  Arms: PC CARES Intervention

SUMMARY:
This participatory, pragmatic efficacy-implementation trial evaluates the impact of Promoting Community Conversations About Research to End Suicide (PC CARES) to evaluate Learning Circle (LC) participant outcomes (AIM#1), community-wide diffusion effects, and efficacy by tracking youth impact (AIM#2), while finding sustainable ways to scale PC CARES to other Alaska Native (AN) communities (AIM#3).

DETAILED DESCRIPTION:
AIM#1 will assess how (and if) our intervention engages the presumed proximal mechanisms of change: personal (self-efficacy) and collective (CoP) resources and skills (including knowledge) as well as distal outcomes (engagement in suicide prevention behaviors) to address suicide in the participants' own community. Using a multilevel growth model, we examine the changes in proximal outcomes of suicide prevention knowledge, self-efficacy, collaborations for a 'community of practice' (CoP), and distal outcomes of prevention-oriented behaviors of adult PC CARES participants (n=250) over time (7 timepoints), testing for moderating effects of dosage (e.g. #LCs attended), community 'readiness'; cross-sector participation on outcomes to inform future PC CARES implementation (AIM#1). Inclusion criteria for participants in Aim#1 are ages 18 and older who participated in PC CARES learning circles.

AIM#2 focuses on diffusion of learning in six randomly selected communities over the same time period as the first aim. The recruitment criteria for participating in this community-wide data collection is to be a resident of the community and age 12 years or older (youth: ages 12-17, and adults: 18 and older). Our community-wide adult and youth measures assess the community-level mechanisms of change (social diffusion), and track youth outcomes. We hypothesize that PC CARES learning circles will encourage adults to develop collaborative relationships within a CoP to implement upstream suicide prevention best practices (SPBPs) in support of youth in their lives. Using community level social network measures, we document the number and type of interactions reported by adults (n=450) over time, capturing social diffusion by comparing the knowledge, self-efficacy, CoP and prevention-oriented behaviors of (1) PC CARES participants, (2) non-participants who are 'close to' participants and (3) others, unrelated to participants (comparison group). In both the Adult and Youth Follow-up Surveys, we characterize closeness (close associates/youth 'close to' participants versus unrelated adults and youth) by asking respondents (Y/N) if they are close to a list of PC CARES participants from their community (i.e. people who attended 4+ LCs). 'Close to' is defined as someone with whom the participant feels closely connected to and interacts with at least weekly.

To assess youth impact (n=300, ages 12-17), we measure youth-reported supportive adult interactions and connectedness (over 7 time points), and pre-post perceived social support, family and community protective factors, comparing outcomes for youth who are 'close to' LC participants versus 'unrelated' youth (comparison group).

AIM#3 combines community-engaged methodologies and evidence-based implementation science frameworks to examine the barriers and enablers of PC CARES implementation in Alaska Native communities. AIM#3 examines implementation outcomes and contextual determinants to further understand how to successfully support community-driven diffusion of SPBPs in extremely rural and remote AN villages. Our evaluation will blend PC CARES' community-engaged approach with two evidence-based and widely used Implementation Science (IS) frameworks (RE-AIM; CFIR 2.0). Using participatory methods, we will sequentially and iteratively seek insights from our community partners, including: Rural Human Service (RHS) Students, RHS instructional teams (Elders; University of Alaska Fairbanks (UAF) Practicum Faculty, mentors), and Community Steering Committee (CSC) members. All RHS student facilitators will be invited to participate in each stage of research, and if interested will be invited to join the Community Steering Committee (CSC). As the RHS student facilitation teams implement LCs as part of their practicum, biweekly zoom/phone calls will support and track RHS student experiences and insights and offer opportunities for peer and mentor support. Monthly written reports will capture each student's community-based actions (e.g., recruitment process, sharing ideas from LCs with the tribal council), their experience of hosting LCs, including 'what worked' (enablers) and implementation barriers. In these various ways, they will reflect on key contextual determinants they are navigating, and how those affect their implementation of PC CARES. Lessons learned or puzzling findings from each of 5 RHS cohorts will be shared with the LSC to gain further insights and to inform the next wave of data collection and analysis. After each wave of implementation, we will conduct focus groups with RHS student facilitators about their overall experience using semi-structured guides informed by our preliminary RE-AIM outcomes (Reach, Effectiveness, Diffusion, Adoption, Implementation and Maintenance). We will transcribe focus groups recordings verbatim and use Dedoose, a qualitative analytic software, for deductive analysis using the RE(D)-AIM construct structure.

ELIGIBILITY:
Inclusion Criteria:

* Anyone aged 12 and over who lives or works in the designated communities may participate in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1075 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Change in Community of Practice (CoP) | Baseline; monthly after each LC, assessed over 5 months; follow-up at 1 month and 6 month after the last LC
  Collaborations for a community of practice (CoP) related to wellness promotion and suicide prevention are measured on a 7-point Agreement Scale (3 survey questions).
  Change in CoP is measured in adult intervention and non-intervention participants.
Change in Suicide Prevention Knowledge | Baseline; monthly after each LC, assessed over 5 months; follow-up at 1 month and 6 month after the last LC
  Knowledge related to suicide prevention are measured using a 7-point Agreement Scale (14 survey questions).
  Suicide prevention knowledge is measured in adult intervention and non-intervention participants.
Change in Self-Efficacy | Baseline; monthly after each LC, assessed over 5 months; follow-up at 1 month and 6 month after the last LC
  Self-efficacy related to wellness promotion and suicide prevention are measured on a 7-point Agreement Scale (5 survey questions).
  Self-efficacy is measured in adult intervention and non-intervention participants.
Change in Youth Connectedness | Baseline; monthly after each LC, assessed over 5 months; and 1 month follow up
  Youth connectedness is measured using a 4-point Agreement Scale (11 survey questions).
  Youth connectedness is measured in youth participants.
Change in Community Protective Factors | Baseline; monthly after each LC, assessed over 5 months; and 1 month follow up
  Community protective factors are measured using a 7-point Agreement Scale (9 survey questions). Community protective factors is measured in youth participants.
Change in Self-Reported Supportive Interactions with Adults | Baseline; monthly after each LC, assessed over 5 months; and 1 month follow up
  Self-reported supportive interactions are measured using a 6-point Frequency Scale (10 survey questions).
  Self-reported supportive interactions are measured in youth participants.
Change in Perceived Social Support | Baseline; monthly after each LC, assessed over 5 months; and 1 month follow up
  Perceived social support is measured using a 7-point Agreement Scale (11 survey questions). Perceived social support is measured in youth participants.
Change in Suicide Prevention-Oriented Behaviors | Baseline; monthly after each LC, assessed over 5 months; follow-up at 1 month and 6 month after the last LC
  Behaviors related to wellness promotion and suicide prevention is measured across four areas: (1) Interpersonal support (9 items); (2) Lethal means reduction (5 items); (3) Postvention (8 items); (4) Working with others to prevent suicide and promote health (19 items). Participants are asked how often they have engaged in these prevention-oriented actions in the last 30 days and with whom using a 7-point frequency scale.
  Suicide prevention-oriented behaviors are measured in adult intervention and non-intervention participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wexler, PhD, Principal Investigator — Univer
Locations (2):
- United States (2):
  - Rural Human Services Program, Fairbanks, Alaska
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No
It is not appropriate for our study and would require additional tribal approvals.

REFERENCES:
- [Background] Markowski KL, White L, Harcey SR, Schmidt T, McEachern D, Habecker P, Wexler L. What Kinds of Support are Alaska Native Youth and Young Adults Reporting? An Examination of Types, Quantities, Sources, and Frequencies of Support. Health Promot Pract. 2023 Sep;24(5):863-872. doi: 10.1177/15248399221115065. Epub 2022 Sep 1. PMID 36047453
- [Background] Wexler L, Rataj S, Ivanich J, Plavin J, Mullany A, Moto R, Kirk T, Goldwater E, Johnson R, Dombrowski K. Community mobilization for rural suicide prevention: Process, learning and behavioral outcomes from Promoting Community Conversations About Research to End Suicide (PC CARES) in Northwest Alaska. Soc Sci Med. 2019 Jul;232:398-407. doi: 10.1016/j.socscimed.2019.05.028. Epub 2019 May 23. PMID 31151026
- [Background] Wells CC, White L, Schmidt T, Rataj S, McEachern D, Wisnieski D, Garnie J, Kirk T, Moto R, Wexler L. Adapting PC CARES to Continue Suicide Prevention in Rural Alaska During the COVID-19 Pandemic: Narrative Overview of an In-Person Community-Based Suicide Prevention Program Moving Online. Am Indian Alsk Native Ment Health Res. 2022;29(2):126-154. doi: 10.5820/aian.2902.2022.126. PMID 35881985
- [Background] Wexler L, McEachern D, DiFulvio G, Smith C, Graham LF, Dombrowski K. Creating a Community of Practice to Prevent Suicide Through Multiple Channels: Describing the Theoretical Foundations and Structured Learning of PC CARES. Int Q Community Health Educ. 2016;36(2):115-22. doi: 10.1177/0272684X16630886. Epub 2016 Feb 15. PMID 26880738
- [Background] Trout L, McEachern D, Mullany A, White L, Wexler L. Decoloniality as a Framework for Indigenous Youth Suicide Prevention Pedagogy: Promoting Community Conversations About Research to End Suicide. Am J Community Psychol. 2018 Dec;62(3-4):396-405. doi: 10.1002/ajcp.12293. PMID 30561803
- [Background] White LA, Wexler L, Weaver A, Moto R, Kirk T, Rataj S, Trout L, McEachern D. Implementation beyond the clinic: Community-driven utilization of research evidence from PC CARES, a suicide prevention program. Am J Community Psychol. 2022 Dec;70(3-4):365-378. doi: 10.1002/ajcp.12609. Epub 2022 Jun 28. PMID 35762450
- See also: Description: Site describing the PC CARES philosophy, curriculum, team, and how people can get involved — http://www.pc-cares.org